CLINICAL TRIAL: NCT03242122
Title: Evaluation of Carbohydrates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BL37 Part 1
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Glycemic Index

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CHO Control 1 Glucose (Active Comparator): 25 g glucose
  Interventions: Other: CHO Control 1 and 2 Glucose
- CHO Experimental 1 Slowly Digested (Experimental): 25 g slowly-digested carbohydrate blend
  Interventions: Other: CHO Experimental 1 Slowly Digested
- CHO Experimental 2 Digestion Resistant (Experimental): 25 g digestion-resistant carbohydrate blend
  Interventions: Other: CHO Experimental 2 Digestion Resistant
- CHO Experimental 3 Low Sugar (Experimental): 25 g low sugar carbohydrate blend
  Interventions: Other: CHO Experimental 3 Low Sugar
- CHO Experimental 4 Maltodextrin (Experimental): 25 g maltodextrin
  Interventions: Other: CHO Experimental 4 Maltodextrin
- CHO Control 2 Glucose (Active Comparator): 25 g glucose
  Interventions: Other: CHO Control 1 and 2 Glucose

INTERVENTIONS:
Other: CHO Control 1 and 2 Glucose — mixed in 237 ml/8 fl oz of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Control 1 Glucose; CHO Control 2 Glucose
Other: CHO Experimental 1 Slowly Digested — mixed in 237 ml/8 fl oz of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 1 Slowly Digested
Other: CHO Experimental 2 Digestion Resistant — mixed in 237 ml/8 fl oz of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 2 Digestion Resistant
Other: CHO Experimental 3 Low Sugar — mixed in 237 ml/8 fl oz of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 3 Low Sugar
Other: CHO Experimental 4 Maltodextrin — mixed in 237 ml/8 fl oz of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 4 Maltodextrin

SUMMARY:
The study is open-label with a randomized, cross-over design using standard Gl methodology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are males or non-pregnant females in good health.
* Subjects must be eligible to receive income in Canada and must demonstrate OHIP or equivalent medical coverage.

Exclusion Criteria:

* Subject with any type of food allergy or with a known history of AIDS, hepatitis, diabetes or a heart condition.
* Subject taking medication, or with any condition which might, in the opinion of the PI either make participation dangerous to the subject or to others or affect the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Blood glucose response curve | 0 to 120 minutes
  area under the curve (AUG)

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (1):
- Glycemic Index Laboratories Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided